CLINICAL TRIAL: NCT05736172
Title: Effect of Therapeutic Education on Pain Levels and Brain Neurotrophic Factor in Patients With Chronic Pain.
Brief Title: 3h of PNE on BDNF and Pain Levels
Acronym: PNE/BDNF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Raúl Ferrer-Peña, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3HPNEBDNF
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: bdnf; pain neuroscience education
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain group education (Experimental): In this group, the education session will be provided in a face-to-face group setting.
  Interventions: Behavioral: Pain neuroscience grupal education
- Pain material education (Active Comparator): In this group the same education session will be provided in written form by means of a leaflet.
  Interventions: Behavioral: Pain neuroscience grupal education

INTERVENTIONS:
Behavioral: Pain neuroscience grupal education — The face to face education group will be carried out with a physiotherapist addressing various topics in the neurosciences of pain. In the active control group, information will only be provided in written form for the individual patient to read.
  Other Names: Pain neuroscience written education

SUMMARY:
The promotion of neuroplasticity in conjunction with strategies for restructuring maladaptive cognitions that largely cause the activation of neural networks that contribute to the perpetuation of pain is therefore a fundamental neurophysiological principle for establishing a neurophysiological basis for pain.

perpetuation of pain, is therefore a fundamental neurophysiological principle for establishing physiotherapy therapeutic to establish therapeutic strategies from physiotherapy that contribute to improve the quality of life of patients with chronic pain. Based on the theory that neurotrophic factors such as BDNF play a fundamental role in the initiation and or maintenance of hyperexcitability of central neurons in pain, we consider that the levels of this neurotrophic factor, such as BDNF, may have an important role in the perpetuation of pain. That the levels of this neurotrophic factor may be modified by the application of a therapeutic education protocol, favoring therapeutic education protocol, favoring a reduction in pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 18 to 65 years with musculoskeletal pain for a minimum of 3 months
* patients recruited by information pamphlets from the university clinic of the Rey Juan Carlos University, and CSEU La Salle
* ability to perform all the clinical tests and to understand the study process, as well as to obtain informed consent.

Exclusion Criteria:

-Systemic, neurological, oncological or inflammatory diseases; psychiatric pathologies, pregnancy, type II diabetes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | three hours
  Pain intensity assessed with the 100 mm Visual Analog Scale, in which the patient is asked about his or her pain level at that moment, with one side being "no pain" and the other extreme being "the worst pain imaginable".
BDNF level | three hours
  BDNF level measured in blood serum by ELISA kit at baseline and at the end of the intervention.

SECONDARY OUTCOMES:
Anxiety and Depression (HADS) | 3 hours
  Anxiety and depression will be assessed using the Spanish validated version of the HADS. The HADS is a selfadministered measure with 14 items in total that ask the client to reflect on their mood in the past week. Seven items assess depression, 5 of which are markers for anhedonia (an inability to experience pleasure), and 2 concern appearance and feelings of slowing down. Seven items assess anxiety, of which 2 assess autonomic anxiety (panic and butterflies in the stomach), and the remaining 5 assess tension and restlessness (Dunbar, Ford, Hunt, & Der, 2000).
Quality of life (EQ-5D) | 3 hours
  The EQ-5D is a generic HRQoL. HRQoL that can be used both in relatively healthy individuals (general population) and in groups of patients with different pathologies.
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem; see appendix).7 8 A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status with 100 indicating the best health status.
Pain Catastrophism Scale (PCS) | 3 hours
  Pain Catastrophism will be measured with the Spanish version of the Pain Catastrophism Scale. The Pain Catastrophizing Scale (PCS) is a 13-item self-report questionnaire considered to be the most frequent and extensively studied tool to assess pain catastrophizing for chronic pain. Good levels of content and construct validity, internal consistency and test-retest reliability of the PCS have been reported in studies examining different musculoskeletal disorders and different language versions.
  The PCS total score is computed by summing responses to all 13 items. PCS total scores range from 0 - 52. The PCS subscales are computed by summing the responses to the following items: Rumination: Sum of items 8, 9, 10, 11 Magnification: Sum of items 6, 7, 13 Helplessness: Sum of items 1, 2, 3, 4, 5, 12
Pain Severity Level (GCPS-R) | 3 hours
  Pain severity will be measured Chronic Pain Grading Scale Description: A measure of pain intensity and interference with normal daily activities. Format: 7 items Scoring: Scores for 6 of the items range from 0 (no pain) to 10 (pain as bad as it could be). The one remaining item requires filling in the number of days that pain has kept respondents from their typical activities.
  Scores classify respondents into one of 4 levels of pain intensity and activity interference:
  Low disability and low pain intensity Low disability and high p

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Di Bonaventura, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Silvia Di Bonaventura, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No